CLINICAL TRIAL: NCT01156675
Title: A Prospective Randomized Clinical Investigation of the FLEXUS(TM) Interspinous Spacer: A Pivotal Study
Brief Title: Study Evaluating the Safety and Effectiveness of the FLEXUS(TM) Interspinous Spacer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Globus Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GPR003
Record Dates: First submitted 2010-07-01; First posted 2010-07-05 (Estimated); Results first posted 2018-04-27 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Back pain; Pain; Spinal Diseases; Spinal Stenosis; Lumbar Vertebrae; Spinal Canal
MeSH Terms: conditions — Spinal Stenosis; Back Pain; Pain; Spinal Diseases

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- FLEXUS™ Interspinous Spacer (Experimental)
  Interventions: Device: FLEXUS(TM) Interspinous Spacer
- XSTOP® Interspinous Spacer (Active Comparator)
  Interventions: Device: XSTOP® Interspinous Spacer

INTERVENTIONS:
Device: FLEXUS(TM) Interspinous Spacer — Treatment of lumbar spinal stenosis with the FLEXUS™ Interspinous Spacer
  Arms: FLEXUS™ Interspinous Spacer
Device: XSTOP® Interspinous Spacer — Treatment of lumbar spinal stenosis with the XSTOP® Spacer
  Arms: XSTOP® Interspinous Spacer

SUMMARY:
The purpose of this investigation is to evaluate the safety and effectiveness of the FLEXUS™ Interspinous Spacer as compared to the XSTOP® Spacer for the treatment of patients who are suffering from lumbar spinal stenosis at one or two contiguous levels.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar spinal stenosis as defined by leg, buttock or groin pain, with or without back pain, that relieves during flexion, with radiographic confirmation of spinal stenosis by CT or MRI scans at one or two contiguous levels between L1 and S1. If back pain is also present, it must be partially relieved during flexion
* Narrowing of the spinal canal, nerve root canal or intervertebral foramen at one or two levels
* Able to sit for 50 minutes without pain
* Able to walk 50 feet or more
* Age 50 years or over
* Has completed at least 6 months of conservative treatment
* Has a Zurich Claudication Questionnaire (ZCQ) score of ≥ 1.5 for Physical Function (PF) and ≥ 1.5 for Symptom Severity (SS)
* Other as specified in the approved protocol

Exclusion Criteria:

* Cannot sit for 50 minutes without pain
* Cannot walk for more than 50 feet
* Unremitting pain in any spinal position
* Axial back pain only without leg, buttock, or groin pain
* Fixed motor deficit
* Cauda equine syndrome, defined as neural compression causing neurogenic bowel (rectal incontinence) or bladder (bladder retension or incontinence) dysfunction
* Severe symptomatic lumbar spinal stenosis at more than two levels
* Significant instability of the lumbar spine
* Has had any surgery of the lumbar spine
* Morbid obesity defined as a body mass index >40 or a weight more than 100 lbs over ideal body weight
* Active systemic disease such as AIDS, HIV, Hepatitis, etc.
* Active systemic or local infection
* Angina, active rheumatoid arthritis, advanced diabetes or any other systemic disease that would affect the subject's welfare or outcome of the study
* Osteoporosis, defined as DEXA bone density measured T-score < -2.5
* Spinal metastasis to the vertebrae
* Known allergy to device materials titanium, tantalum, or polyetheretherketone (PEEK) polymer
* Other as specified in approved protocol

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2008-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Skyridge Medical Center, Denver, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- X-STOP® Interspinous Spacer: X-STOP® Interspinous Spacer: Treatment of lumbar spinal stenosis with the XSTOP® Spacer
- No Treatment: Not treated with FLEXUS or X-STOP
Period: Overall Study
Arm/Group | FLEXUS™ Interspinous Spacer | X-STOP® Interspinous Spacer | No Treatment
Started | 107 | 106 | 2
Completed | 73 | 81 | 0
Not Completed | 34 | 25 | 2
Not completed — Death | 5 | 3 | 0
Not completed — No data | 29 | 22 | 2

BASELINE CHARACTERISTICS:
Groups:
- X-STOP® Interspinous Spacer: X-STOP® Interspinous Spacer: Treatment of lumbar spinal stenosis with the X-STOP® Spacer
- Total: Total of all reporting groups
Arm/Group | FLEXUS™ Interspinous Spacer | X-STOP® Interspinous Spacer | No Treatment | Total
Number analyzed (Participants) | 107 | 106 | 2 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (8.93) | 67.3 (8.88) | 71.5 (4.95) | 67.8 (8.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 46 | 1 | 101
  Male | 53 | 60 | 1 | 114
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 98 | 102 | 2 | 202
  Race: Black | 7 | 3 | 0 | 10
  Race: Asian | 1 | 0 | 0 | 1
  Race: Hispanic | 1 | 0 | 0 | 1
  Race: Other | 0 | 1 | 0 | 1
Weight (lbs) [Mean (Standard Deviation); unit: lbs] | 181.8 (33.87) | 193.2 (37.75) | 195.0 (77.78) | 187.5 (36.45)
Height (inches) [Mean (Standard Deviation); unit: inches] | 67.0 (3.62) | 67.2 (3.94) | 66.0 (11.31) | 67.1 (3.84)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Less Pain/Disability Using the Zurich Claudication Questionnaire (ZCQ) Score
Description: Change in the Zurich Claudication Questionnaire (ZCQ) score at 24 months compared with the score at baseline as follows:
  * Change of >0.5 points in Physical Function on a scale of 1-4 points (lower values are considered a better outcome)
  * Change of >0.5 points in Symptom Severity on a scale of 1-5 points (lower values are considered a better outcome)
  * Satisfaction of <2.5 points on a scale of 1-4 points (lower values are considered a better outcome) The Zurich Claudication Questionnaire is a three part form that quantifies severity of symptoms, physical function characteristics, and patient's satisfaction after treatment.
Time Frame: 24 months
Population: The Overall Number of Participants Analyzed is not consistent with numbers provided in the Participant Flow module. The discrepancy in the numbers is due to an additional subject having ZCQ data at 24 months in the FLEXUS arm and one less subject with ZCQ data at 24 months in the X-STOP group. No data was collected for the "No Treatment" arm.
Measure: Count of Participants; unit: Participants
Arm/Group | FLEXUS™ Interspinous Spacer | X-STOP® Interspinous Spacer | No Treatment
Number analyzed (Participants) | 74 | 80 | 0
Participants | 42 | 50 | 0

2. Primary Outcome: Number of Participants With a Successful Neurologic Status
Description: Neurological status is based on four types of measurement parameters: motor, sensory, reflexes, and special assessments. Each parameter will be coded as follows:
  Motor 0 Total Paralysis
  1. Palpable or Visible Contraction
  2. Active Movement, Gravity Eliminated
  3. Active Movement, Against Gravity
  4. Active Movement, Against Some Resistance
  5. Active Movement, Against Full Resistance
  Sensory 0 Absent
  1. Impaired
  2. Normal
  Reflexes 0 Absent or Trace
  1. Hyper-reflexic
  2. Normal or hypo-reflexic
  Straight Leg Raise 0 0°-70° (abnormal)
  1 >70°-90° (normal)
  If all evaluations for the parameter are determined to be normal, then the parameter is given a normal status. If any evaluations for the parameter are abnormal, then the parameter is given an abnormal status. The overall neurological status will be considered a success if and only if all the four parameters are stable or improved.
Time Frame: 24 months
Population: The Overall Number of Participants Analyzed is not consistent with numbers in the Participant Flow module. The discrepancy is due to two less subjects having neurologic status data at 24 months in the FLEXUS arm and one less subject with neurologic status data at 24 months in the X-STOP arm. No data was collected for the "No Treatment" arm.
Measure: Count of Participants; unit: Participants
Arm/Group | FLEXUS™ Interspinous Spacer | X-STOP® Interspinous Spacer | No Treatment
Number analyzed (Participants) | 71 | 80 | 0
Participants | 60 | 69 | 0

3. Primary Outcome: Number of Participants With no Additional Surgery for Lumbar Spinal Stenosis at the Spinal Level That Was Treated
Description: Measures the number of participants who did not have another surgery for treatment of lumbar spinal stenosis at the same spinal level that was originally treated. Data, including adverse events, were monitored, evaluated and assessed for evidence of additional surgical treatment at the spinal level that was originally treated.
Time Frame: 24 months
Population: The Overall Number of Participants Analyzed in the FLEXUS arm and X-STOP arm is the number of subjects who started the Study in the respective arm. No data was collected for the "No Treatment" arm.
Measure: Count of Participants; unit: Participants
Arm/Group | FLEXUS™ Interspinous Spacer | X-STOP® Interspinous Spacer | No Treatment
Number analyzed (Participants) | 107 | 106 | 0
Participants | 90 | 99 | 0

4. Primary Outcome: Number of Participants With an Absence of Implant-related Complications
Description: Absence of implant-related complications, including device dislodgement, defined as:
  * Failure of implant material (e.g. fracture);
  * Implant migration outside of the interspinous space (posteriorly beyond the posterior margin of the spinous processes, anteriorly within the spinal canal, or laterally more than half of the implant width); or
  * Other complications that can be specifically associated with the implanted device.
Time Frame: 24 months
Population: The Overall Number of Participants Analyzed in the FLEXUS arm and X-STOP arm is the number of subjects who started the Study in the respective arms. No data was collected for the "No Treatment" arm.
Measure: Count of Participants; unit: Participants
Arm/Group | FLEXUS™ Interspinous Spacer | X-STOP® Interspinous Spacer | No Treatment
Number analyzed (Participants) | 107 | 106 | 0
Participants | 84 | 97 | 0

5. Secondary Outcome: Mean Oswestry Disability Index (ODI) at 24 Months
Description: The Oswestry Disability Index (ODI) questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each topic is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The subject chooses the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. Scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability.
Time Frame: 24 months
Population: The Overall Number of Participants Analyzed is not consistent with numbers in the Participant Flow module. The discrepancy is due to ten less subjects having ODI data at 24 months in the FLEXUS arm and four less subject with ODI data at 24 months in the X-STOP arm. No data was collected for the "No Treatment" arm.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | FLEXUS™ Interspinous Spacer | X-STOP® Interspinous Spacer | No Treatment
Number analyzed (Participants) | 63 | 77 | 0
score | 19.2 (17.97) | 17.4 (14.15) |

6. Secondary Outcome: Mean Visual Analog Scale (VAS) - Back Pain at 24 Months
Description: The visual analog scale (VAS) is a questionnaire used to quantify a subjective experience, such as the intensity of pain. The scale is a 100mm line labeled with "no pain" on the left border and "as severe as it could be" on the right border. The subject is instructed to make a mark along the line to represent the intensity of back pain currently being experienced; 0mm is equal to no pain and 100mm is pain as severe as it could be. The clinician records the distance of the mark in millimeters from the left end of the scale.
Time Frame: 24 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | FLEXUS™ Interspinous Spacer | X-STOP® Interspinous Spacer | No Treatment
Number analyzed (Participants) | 62 | 77 | 0
millimeters | 20.2 (27.77) | 18.8 (27.36) |

7. Secondary Outcome: Mean Visual Analog Scale (VAS) - Right Leg Pain at 24 Months
Description: The visual analog scale (VAS) is a questionnaire used to quantify a subjective experience, such as the intensity of pain. The scale is a 100mm line labeled with "no pain" on the left border and "as severe as it could be" on the right border. The subject is instructed to make a mark along the line to represent the intensity of right leg pain currently being experienced; 0mm is equal to no pain and 100mm is pain as severe as it could be. The clinician records the distance of the mark in millimeters from the left end of the scale.
Time Frame: 24 months
Population: The Overall Number of Participants Analyzed is not consistent with numbers in the Participant Flow module. The discrepancy is due to eleven less subjects having VAS data at 24 months in the FLEXUS arm and four less subject with VAS data at 24 months in the X-STOP arm. No data was collected for the "No Treatment" arm.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | FLEXUS™ Interspinous Spacer | X-STOP® Interspinous Spacer | No Treatment
Number analyzed (Participants) | 62 | 77 | 0
millimeters | 16.2 (26.72) | 9.2 (15.77) |

8. Secondary Outcome: Mean Visual Analog Scale (VAS) - Left Leg Pain at 24 Months
Description: The visual analog scale (VAS) is a questionnaire used to quantify a subjective experience, such as the intensity of pain. The scale is a 100mm line labeled with "no pain" on the left border and "as severe as it could be" on the right border. The subject is instructed to make a mark along the line to represent the intensity of left leg pain currently being experienced; 0mm is equal to no pain and 100mm is pain as severe as it could be. The clinician records the distance of the mark in millimeters from the left end of the scale.
Time Frame: 24 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | FLEXUS™ Interspinous Spacer | XSTOP® Interspinous Spacer | No Treatment
Number analyzed (Participants) | 62 | 77 | 0
millimeters | 13.2 (27.43) | 10.7 (20.11) |

9. Secondary Outcome: Change of Quality of Life
Description: Change in mental or physical composite score of the short form SF36
Time Frame: 24 months
Population: The short form SF36 was administered to study patients; however, we do not have the proprietary scoring system. Hence the scores could not be calculated.
Arm/Group | FLEXUS™ Interspinous Spacer | X-STOP® Interspinous Spacer | No Treatment
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: Adverse events were reviewed and classified by a Clinical Events Committee (CEC).
Arm/Group | FLEXUS™ Interspinous Spacer | X-STOP® Interspinous Spacer | No Treatment
All-Cause Mortality (participants affected / at risk) | 5/107 | 3/106 | 0/2
Serious Adverse Events (participants affected / at risk) | 41/107 | 28/106 | 0/2
Other Adverse Events (participants affected / at risk) | 77/107 | 72/106 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FLEXUS™ Interspinous Spacer (N=107) | X-STOP® Interspinous Spacer (N=106) | No Treatment (N=2)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Cardiovascular (Cardiac disorders) | 8 | 5 | 0
Carpal Tunnel Syndrome (General disorders) | 1 | 0 | 0
Cerebrovascular (Vascular disorders) | 2 | 0 | 0
Compressive Peripheral Neuropathy (Non-CTS) (Nervous system disorders) | 0 | 1 | 0
Death (General disorders) | 5 | 3 | 0
Gastrointestinal (Gastrointestinal disorders) | 2 | 1 | 0
Infection - Superficial Wound (Infections and infestations) | 0 | 1 | 0
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Other (General disorders) | 1 | 0 | 0
Pain - Back (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain - Hip (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0
Pain - Lower Extremities (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Pain - Neck and/or Upper Extremities (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Pseudoarthrosis (General disorders) | 1 | 0 | 0
Surgery - Index Level (Surgical and medical procedures) | 21 | 12 | 0
Surgery - Non-Index Lumbar (Surgical and medical procedures) | 3 | 0 | 0
Surgery - Non-Index Lumbar (Surgical and medical procedures) | 1 | 0 | 0
Trauma (Social circumstances) | 1 | 0 | 0
Urogenital (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FLEXUS™ Interspinous Spacer (N=107) | X-STOP® Interspinous Spacer (N=106) | No Treatment (N=2)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Cardiovascular (Cardiac disorders) | 6 | 3 | 0
Carpal Tunnel Syndrome (CTS) (General disorders) | 0 | 1 | 0
Dysesthesia - Lower Extremities (Nervous system disorders) | 1 | 2 | 0
Gastrointestinal (Gastrointestinal disorders) | 2 | 4 | 0
Headache (General disorders) | 3 | 1 | 0
Infection - Other (Infections and infestations) | 6 | 1 | 0
Infection - Superficial Wound (Infections and infestations) | 2 | 5 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Neurological (Nervous system disorders) | 0 | 4 | 0
Other (General disorders) | 10 | 6 | 0
Pain - Back (Musculoskeletal and connective tissue disorders) | 34 | 32 | 1
Pain - Back and Hip (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Pain - Back and Lower Extemities (Musculoskeletal and connective tissue disorders) | 11 | 9 | 0
Pain - Hip (Musculoskeletal and connective tissue disorders) | 12 | 9 | 0
Pain - Lower Extremities (Musculoskeletal and connective tissue disorders) | 26 | 33 | 1
Pain - Lower Extremities with Dysesthesia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
Pain - Neck and/or Upper Extremities (Musculoskeletal and connective tissue disorders) | 12 | 8 | 0
Pain - Other (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Paresthesia - Lower Extremities (General disorders) | 11 | 10 | 0
Paresthesia - Upper Extremities (General disorders) | 2 | 1 | 0
Psychological (Psychiatric disorders) | 2 | 0 | 0
Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Spinous Process Fracture (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Surgery - Index Level (General disorders) | 1 | 0 | 0
Trauma (Social circumstances) | 6 | 3 | 0
Urogenital (Renal and urinary disorders) | 3 | 2 | 0
Weakness (General disorders) | 3 | 3 | 0
Wound Issue (Injury, poisoning and procedural complications) | 1 | 3 | 0
Pain - Back and Lower Extemities with Dysesthesia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No